CLINICAL TRIAL: NCT05555628
Title: Comparison of Two Exercise Therapy Protocols in Patients With Bruxism: A Randomized Controlled Trial
Brief Title: Comparison of Two Exercise Therapy Protocols in Patients With Bruxism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, GulOznur KARABICAK, Phd PT Principal Investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 92340882-050.04.04
Record Dates: First submitted 2022-08-26; First posted 2022-09-27 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Bruxism
Keywords: bruxism; physiotherapy; exercise therapy; occlusal splint; pain; rehabilitation
MeSH Terms: conditions — Bruxism; Pain

STUDY DESIGN:
Intervention Model Description: Patients in Groups I and II will be included in an exercise program that will last for 45 minutes, two days a week, for 6 weeks. All treatments will be carried out by a physiotherapist with more than 10 years of experience in the field. The patients will be treated independently from each other. The treatment protocols of the patients in exercise therapy group will be revised with 2-week controls, and their progress will be followed up with new exercises. Patients who do not come to two consequtive treatments to the treatment protocol will be excluded from the study.
  Occlusal Splint Group; It will consist of two separate sessions, one week apart. It is aimed to eliminate possible incompatibilities by calling the patients for the control one week after the splints are delivered.
  Assessments will be performed three times: prior to group assignment (baseline), immediately after the end of the treatment (week 6), and at the control of the 12th week.
Who Masked: Outcomes Assessor
Masking Description: Patients eligible to participate in the study will be assessed by a researcher who is blind to group assignment. The assessor will only see the patients during the evaluation. In this way, the masking of group assignment will be ensured.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mandibular Exercise (Experimental): At the beginning of the treatment, the therapist will perform a soft tissue massage to the patient's muscles. Then, an exercise protocol for specific muscles (masseter, temporal muscles, mandibular region muscles) will be administered. This group, the exercise will focus only on the chin area, not general like posture.
  Interventions: Other: Mandibular Exercise
- Mandibular and Postural Exercise (Experimental): The patients will perform posture exercises, including stabilization of the upper body and cervical region, accompanied by a physiotherapist. A theraband suitable for the patient's muscular strength will be used for posture exercises,. The appropriate therabant selection will be decided by a maximum repetition method.
  Interventions: Other: Mandibular Exercise; Other: Mandibular Exercise and Postural Exercise Group
- Occlusal Splint (Active Comparator): The patients assigned to this group will be treated by the occlusal splint administered by the dentist and the recommendations that they should pay attention to in daily life.
  Occlusal splints will be prepared according to previously published criteria by Okeson and other researchers. Occlusal splint measurement and production will be done by technicians with 5 years of experience. Using the models obtained from the maxillary measurements of the patients, 0.5 mm thick thermoplastic rigid splints will be prepared and adjusted according to the patient's occlusion. Occlusal splints will be prepared for night use only. Patients will use splints every night for 6 weeks. Splint use of the patients and possible side effects or plaque-related disorders will be followed up with phone calls to be made every 2 weeks.
  Interventions: Other: Occlusal Splint Group

INTERVENTIONS:
Other: Mandibular Exercise — Patients will receive exercise treatment twice weekly for 6 weeks period. Every session will last approximately 40 minutes
  Arms: Mandibular Exercise; Mandibular and Postural Exercise
Other: Mandibular Exercise and Postural Exercise Group — Patients will receive exercise treatment twice weekly for 6 weeks period. Every session will last approximately 40 minutes
  Arms: Mandibular and Postural Exercise
Other: Occlusal Splint Group — Patients will use occlusal splints for 6 weeks. The occlusal splints will be used only sleep time.
  Arms: Occlusal Splint

SUMMARY:
The main purpose of this planned research is to investigate the effectiveness of three different methods used for the treatment of bruxism. Two of these are physiotherapy-specific exercise treatment protocols (1.posture and proprioception exercises 2. Jaw area strengthening exercises) and a control group, (occlusal splint therapy) will take place during the study.

DETAILED DESCRIPTION:
The current study is planned as a parallel group, randomized controlled trial. Patients who apply to Adnan Menderes University Faculty of Dentistry between June 2022 and January 2023 and diagnosed with bruxism after the examination will be screened for the study. Aydın Adnan Menderes University Faculty of Dentistry is a hospital that serves an average of 400 patients per day.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of sleep Bruxism according to the criteria of the International Classification of Sleep Disorders (ICSD) of the American Academy of Sleep Medicine (AASM) (5);
2. 18-50 age range
3. The diagnosis of awake bruxism, which was determined by a positive answer to the questions of the questionnaire developed according to Pintado's recommendations (6);
4. Pain around the jaw is 3 or more on the visual analog scale (7)
5. Patients who volunteered to participate in the study

Exclusion Criteria:

1. Systemic and/or degenerative disorders
2. Neurological or psychiatric diseases (excluding anxiety and depression)
3. Use of drugs that affect sleep or motor behavior
4. Arthrogenic or mixed temporomandibular disorder
5. Axis I myogenic TMD according to investigational diagnostic criteria for temporomandibular disorders (RDC/TMD)
6. Patients using total prosthesis
7. Direct trauma or previous surgical intervention in the orofacial region
8. Patients using muscle relaxants and non-steroidal anti-inflammatory drugs.
9. Patients using removable prostheses
10. Patients who have received any treatment for bruxism
11. Patients who did not want to participate in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 21 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Mandibular Motion | baseline, 6 week, 12 week
  change in active mouth opening, lateral jaw movements and protrusion of mandible
Change in Pain level: pain intensity via Visual Analog Scale | baseline, 6 week, 12 week
  Visual analog scale will be used for the change in pain severity. In a straight line adjusted to 10 cm, the patient is asked to mark the intensity of pain felt at the moment on jaw area. A value of 0 is used to describe the absence of pain, and a value of 10 to describe an unbearable pain. Patients will be asked to rate their pain at the time of assessment (not in the past week or month).
Change in Pain level: pain threshold. | baseline, 6 week, 12 week
  Pressure algometry will be used to assess the pain threshold. This device, which has a pressure area of 1 cm in diameter, shows the applied pressure objectively. The pressure algometer, will be applied by pressing the patient's trigger points (masseter, temporal, trapezius muscles) at an angle of 90 degrees, is calculated by recording the pressure that occurs when the person expresses that he/she feels the pain for the first time. The patient will be positioned seated. The average of the three measurement results to be made is recorded as an evaluation.

SECONDARY OUTCOMES:
The Pittsburg Sleep Quality Index was used to assess sleep quality. | baseline, 6 week, 12 week
  The Pittsburg Sleep Quality Index was developed by Buysse et al. (1989) to evaluate sleep quality in psychiatry practices and clinical studies (1). The items in the PUKI were arranged using clinical observations of patients with sleep disorders, other scales related to sleep quality mentioned in the literature, and an 18-month clinical observation period related to The Pittsburg Sleep Quality Index. The Turkish validity and reliability study of this scale was carried out by Ağargün (1996) (2). The total score of the questionnaire ranges between 0 to 21. 5 points and more refers to bad sleep quality
Oral Behaviours Checklist questionnaire was used to examine the oral habits of of the participants. | baseline, 6 week, 12 week
  The questionnaire, which questions how often parafunctional habits such as clenching, grinding, nail, lip, cheek, pencil biting, gum chewing have been done in the last month, is answered with a 4-point Likert scale. The total score of the the Oral Behaviours Checklist will be used for the analyses. A person's overall score can range from 0 to 84. The validity and reliability of the questionnaire has been demonstrated within the scope of the RDC/TMD Validation project (3).
Postural alterations of the patients will be assessed by using the photographic method. | baseline, 6 week, 12 week
  Within the scope of the evaluation, craniovertebral and craniocervical angles will be evaluated. For this purpose, an silence environment where the patients are comfortable will be provided, and photographs will be taken from the same lateral direction with the help of a camera located on a triple stand 1.5m away, fixed at a height of 115cm. All necessary procedure explanations are available in the relevant resource (4). With this method, an objective numerical data is obtained for the evaluation of cervical posture.

CONTACTS AND LOCATIONS:
Overall Officials: Gul Karabicak, PhD, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Adnan Menderes University Faculty of Dentistry, Aydin, Turkey (Türkiye)

REFERENCES:
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Ağargün, M.Y., Kara, H., Anlar, Ö. (1996). The validity and reliability of the Pittsburgh Sleep Quality Index. Türk Psikiyatri Dergisi, 7 (2), 107-115.
- [Background] Markiewicz MR, Ohrbach R, McCall WD Jr. Oral behaviors checklist: reliability of performance in targeted waking-state behaviors. J Orofac Pain. 2006 Fall;20(4):306-16. PMID 17190029
- [Background] Hazar Z, Karabicak GO, Tiftikci U. Reliability of photographic posture analysis of adolescents. J Phys Ther Sci. 2015 Oct;27(10):3123-6. doi: 10.1589/jpts.27.3123. Epub 2015 Oct 30. PMID 26644658
- [Background] American Sleep Disorders Association. The International Classification of Sleep Disorders, Revised: Diagnostic and Coding Manual. Westchester, IL: American Academy of Sleep Medicine; 2005.
- [Background] Pintado MR, Anderson GC, DeLong R, Douglas WH. Variation in tooth wear in young adults over a two-year period. J Prosthet Dent. 1997 Mar;77(3):313-20. doi: 10.1016/s0022-3913(97)70189-6. PMID 9069087
- [Background] Boonstra AM, Schiphorst Preuper HR, Reneman MF, Posthumus JB, Stewart RE. Reliability and validity of the visual analogue scale for disability in patients with chronic musculoskeletal pain. Int J Rehabil Res. 2008 Jun;31(2):165-9. doi: 10.1097/MRR.0b013e3282fc0f93. PMID 18467932
- [Derived] Karabicak GO, Alkan Demetoglu G, Ozkan G, Gunaydin G, Onal Aykar S, Gunaydin OE. Jaw Exercise Versus Jaw & Posture Exercise Therapies in Comparison to Occlusal Splint Effectiveness in Probable Sleep Bruxism: A Randomised Controlled Study. J Oral Rehabil. 2025 Oct;52(10):1629-1640. doi: 10.1111/joor.14027. Epub 2025 May 14. PMID 40369740